CLINICAL TRIAL: NCT01406561
Title: A Randomized, Double-Blind, Parallel Group, Vehicle-Controlled Study to Evaluate the Safety and Efficacy of OMS103HP-S Administered in Joint Irrigation Solution to Subjects Undergoing Arthroscopic Meniscectomy
Brief Title: Safety and Efficacy of OMS103HP-S Administered in Joint Irrigation Solution to Subjects Undergoing Arthroscopic Meniscectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMS103-MEN-002
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Meniscal Tear
Keywords: Meniscectomy; Knee Pain; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMS103HP-S (Experimental): OMS103HP-S injected into vehicle irrigation solution for administration during meniscectomy surgery
  Interventions: Drug: OMS103HP-S
- Vehicle Irrigation Solution (Placebo Comparator): Vehicle Irrigation Solution
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: OMS103HP-S — Proprietary concentration and formulation of OMS103HP in solution (OMS103HP-S) for injection into each 3 liter vehicle irrigation solution bag for use during meniscectomy surgery
  Arms: OMS103HP-S
Drug: Vehicle — 3 Liter bags of vehicle irrigation solution for use during meniscectomy surgery
  Arms: Vehicle Irrigation Solution

SUMMARY:
The purpose of this study is to assess the effect of OMS103HP solution for Injection (OMS103HP-S) and function as measured by the Knee Osteoarthritis Outcome Survey (KOOS) Symptoms subscale through Day 30 compared with vehicle irrigation solution for knee symptoms in subjects undergoing meniscectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent in accordance with governing Institutional Review Board (IRB)/Independent Ethics Committee (IEC) requirements, local regulations, and Health Insurance Portability and Accountability Act (HIPAA) Authorization (or equivalent if locally applicable)
2. In the opinion of the Investigator are able to comply with study-required visits and procedures
3. 18 to 75 years of age, inclusive at the time of screening
4. Have a traumatic or degenerative meniscal cartilage injury (full thickness tear) that occurred at least 14 days prior to the day of arthroscopic surgery that is demonstrated on MRI
5. Planning to undergo unilateral arthroscopic meniscectomy
6. If female and of childbearing potential (i.e., not surgically sterilized or post-menopausal for longer than one year), agree to use a medically accepted method of birth control for the duration of her study involvement
7. At minimal risk from anesthesia and classified according to the American Society of Anesthesiologists Physical Status Classification as either PS-1 (a normal healthy patient) or PS-2 (a patient with mild systemic disease that results in no functional limitation) as determined by the Investigator.

Exclusion Criteria:

1. Significant arthritis in the surgical knee (Grade 3 or 4 on the Kellgren- Lawrence Grading Scale).
2. History of reactive synovial disease
3. History of a complex regional pain syndrome (Type I, i.e., reflex sympathetic dystrophy, or Type II, i.e., causalgia), chronic pain, attendance at a chronic pain clinic, or neurologic disorder associated with sensory deficit of the lower extremities
4. History of fibromyalgia
5. Expected to undergo any of the following procedures concurrent with the meniscectomy:

   * Meniscal repair procedure
   * Patellar tendon debridement
   * Patellar realignment
   * Lateral or retinacular release
   * Excision synovectomy (minor synovectomy to improve arthroscopic visualization is allowed)
   * Concurrent ligamentous procedure
   * Abrasion chondroplasty involving bone
   * Microfracture
   * Chondral transplantation
   * Use of more than three portals
6. Known allergies to any of the individual ingredients in OMS103HP-S, other NSAIDs, aspirin, tricyclic antidepressants, or opioid analgesics
7. Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study
8. Have a job-related claim(s) under dispute or mediation
9. History of drug or alcohol abuse
10. Treatment with an investigational drug or device within 30 days prior to the day of surgery
11. A clinically significant medical condition that in the opinion of the Investigator would put the subject at increased risk, impair the subject's ability to comply with the requirements of the protocol, or confound the interpretation of the data
12. Expected to receive a regional block for analgesia for this procedure
13. Considered by the Investigator for any reason to be an unsuitable candidate for receipt of an investigational drug
14. The Investigator, employee of the investigative site, and/or part of the Investigator/employee's immediate families (defined as current spouse or partner, parent, natural or legally adopted child, stepchild living in the household, grandparent, or grandchild).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
KOOS Symptoms Subscale | 30 days
  To evaluate the effect of OMS103HP-S compared to vehicle when administered in joint irrigation fluid during arthroscopic meniscectomy on knee symptoms as measured by the KOOS Symptoms subscale through Day 30.
Safety | 90 days
  To evaluate the safety of OMS103HP-S compared to vehicle when administered in joint irrigation fluid during arthroscopic meniscectomy on safety as measured by adverse events.

SECONDARY OUTCOMES:
Knee Function in Sport Active patients | 30 Days
  To evaluate the effect of OMS103HP-S compared to vehicle when administered in joint irrigation fluid during arthroscopic meniscectomy on knee function as measured by the KOOS Sports and Recreation subscale through Day 30 in the subset of subjects who participate in sports.
Knee Pain | 30 days
  To evaluate the effect of OMS103HP-S compared to vehicle when administered in joint irrigation fluid during arthroscopic meniscectomy on knee pain as measured by the KOOS Pain subscale through Day 30.
Quality of Life | 30 days
  To evaluate the effect of OMS103HP-S compared to vehicle when administered in joint irrigation fluid during arthroscopic meniscectomy on knee quality of life as measured by the KOOS Quality of Life subscale through Day 30.
Knee Function | 30 days
  To evaluate the effect of OMS103HP-S compared to vehicle when administered in joint irrigation fluid during arthroscopic meniscectomy on knee function as measured by the KOOS Activities of Daily Living subscale through Day 30.
Postoperative Knee Pain | Day of Surgery (day 1)
  To evaluate the effect of OMS103HP-S compared to vehicle when administered in joint irrigation fluid during arthroscopic meniscectomy on postoperative knee pain as measured by the Visual Analog Scale during the day of surgery.
Passive Flexion | 7 Days
  To evaluate the effect of OMS103HP-S compared to vehicle when administered in joint irrigation fluid during arthroscopic meniscectomy on Passive flexion on Day 7.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Whitaker, MD, Study Director — Omeros Corporation
Locations (17):
- United States (17):
  - Orthopedic Surgery Center, Phoenix, Arizona
  - Orthopedic Surgery Center, Tucson, Arizona
  - Orthopedic Surgery Center, Encinitas, California
  - Orthopedic Surgery Center, Laguna Hills, California
  - Orthopedic Surgery Center, Los Angeles, California
  - Orthopedic Surgery Center, Chicago, Illinois
  - Orthopedic Surgery Center, Royal Oaks, Michigan
  - Orthopedic Surgery Center, Bloomington, Minnesota
  - Orthopedic Surgery Center, Edina, Minnesota
  - Orthopedic Surgery Center, New York, New York
  - Orthopedic Surgery Center, The Bronx, New York
  - Orthopedic Surgery Center, Durham, North Carolina
  - Orthopedic Surgery Center, Columbus, Ohio
  - Orthopedic Surgery Center, Altoona, Pennsylvania
  - Orthopedic Surgery Center, State College, Pennsylvania
  - Orthopedic Surgery Center, San Antonio, Texas
  - Orthopedic Surgery Center, Seattle, Washington